CLINICAL TRIAL: NCT06315387
Title: Open Study of Safety, Tolerability and Pharmacokinetic Parameters of Increasing Doses of 4-MUST, Tablets, 128 mg (Valenta Pharm JSC) During Single and Subsequent Multiple Oral Administration in Healthy Volunteers.
Brief Title: Safety, Tolerability and Pharmacokinetics of 4-MUST, Tablets, 128 mg (Valenta Pharm JSC) During Single and Multiple Oral Administration in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: GIB-01-01-2023
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4-MUST, 128 mg (Experimental): Single dose: 1 tablet (128 mg). Multiple dose: 1 tablet (128 mg) 3 times a day for 3 days (first dose on an empty stomach, second and third two hours after meals), once in the morning on an empty stomach on day 4.
  Interventions: Drug: 4-MUST, 1 tablet
- 4-MUST, 256 mg (Experimental): Single dose: 2 tablets (256 mg). Multiple dose: 2 tablets (256 mg) 3 times a day for 3 days (the first intake of the drug on an empty stomach, the second and third - two hours after a meal), once in the morning on an empty stomach on the 4th day.
  Interventions: Drug: 4-MUST, 2 tablets
- 4-MUST, 384 mg (Experimental): Single dose: 3 tablets (384 mg). Multiple dose: 3 tablets (384 mg) 3 times a day for 3 days (the first intake of the drug on an empty stomach, the second and third - two hours after a meal), once in the morning on an empty stomach on the 4th day.
  Interventions: Drug: 4-MUST, 3 tablets

INTERVENTIONS:
Drug: 4-MUST, 1 tablet — 4-methylumbelliferyl trimebutine sulfate, 128 mg
  Arms: 4-MUST, 128 mg
Drug: 4-MUST, 2 tablets — 4-methylumbelliferyl trimebutine sulfate, 256 mg
  Arms: 4-MUST, 256 mg
Drug: 4-MUST, 3 tablets — 4-methylumbelliferyl trimebutine sulfate, 384 mg
  Arms: 4-MUST, 384 mg

SUMMARY:
Study of safety, tolerability and pharmacokinetic parameters of different doses of 4-MUST, tablets, 128 mg (Valenta Pharm JSC) in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and handwritten informed consent form signed by a healthy volunteer to participate in the study prior to any of the study procedures;
2. Males and females between the ages of 18 and 45 years (inclusive) of Caucasian race;
3. Verified diagnosis of "healthy" (absence of abnormalities according to the data of clinical, laboratory, instrumental methods of examination stipulated by the protocol);
4. Blood pressure (BP) level: systolic blood pressure (SBP) from 99 to 129 mmHg (inclusive), diastolic blood pressure (DBP) from 70 to 89 mmHg (inclusive);
5. Heart rate (HR) from 60 to 89 beats/min (inclusive);
6. Respiratory rate (RR) from 12 to 20 per 1 minute (inclusive);
7. Body temperature between 36.0°C and 36.9°C (inclusive);
8. Body mass index (BMI) of 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2, with body mass ≥ 55 kg for males and ≥ 45 kg for females;
9. Agreement to use adequate contraceptive methods throughout the study and for 30 days after completion of the study, for women of preserved reproductive potential, a negative urine pregnancy test result.

Non-inclusion Criteria:

1. Aggravated allergic history;
2. Hypersensitivity to gimecromone and trimebutine and/or excipients included in the investigational medicinal product in anamnesis;
3. Drug intolerance to hymecromone and trimebutine and/or excipients included in the investigational medicinal product in the anamnesis;
4. Hereditary galactose intolerance, lactase deficiency or glucose-galactose malabsorption in the anamnesis;
5. Chronic diseases of the kidney, liver, gastrointestinal tract (GIT), cardiovascular, lymphatic, respiratory, nervous, endocrine, musculoskeletal, genitourinary and immune systems, as well as skin, hematopoietic and visual organs;
6. A history of GIT surgery (except for appendectomy at least 1 year prior to screening);
7. Diseases/conditions that, in the opinion of the investigator, may affect the absorption, distribution, metabolism, or excretion of the investigational drug (ID);
8. Acute infectious diseases less than 4 weeks prior to screening;
9. Taking drugs that have a significant effect on hemodynamics and drugs that affect liver function (barbiturates, omeprazole, cimetidine, etc.) less than 2 months before screening;
10. Regular intake of a medication less than 2 weeks prior to screening and a single intake of a medication less than 7 days prior to screening (including over-the-counter medications, vitamins, supplements, herbs);
11. Blood or plasma donation less than 3 months prior to screening;
12. Use of hormonal contraceptives (in women) less than 2 months prior to screening;
13. Use of depot injections of any medication less than 3 months prior to screening;
14. Pregnancy or lactation period; positive urine pregnancy test for women of preserved reproductive potential;
15. Women with preserved reproductive potential who have a history of unprotected sexual intercourse within 30 days prior to study medication with an unsterilized partner;
16. Participation in another clinical trial less than 3 months prior to screening or concurrent with the present study;
17. Consumption of more than 10 units of alcohol (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of wine, or 50 ml of spirits) per week in the last month prior to study inclusion or history of alcoholism, drug abuse, or medication abuse;
18. Smoking more than 10 cigarettes per day currently, or history of smoking the specified number of cigarettes in the 6 months preceding screening; failure to agree to abstain from smoking for the duration of the hospital stay;
19. Consumption of alcohol, caffeine, and xanthine-containing products in the 7 days prior to taking the study drug;
20. Consumption of citrus fruits, cranberries, rose hips and products containing them, preparations or products containing St. John's wort - 7 days before taking the study drug;
21. Dehydration due to diarrhea, vomiting or other cause within the last 24 hours before taking the study drug;
22. Positive blood test result for antibodies to human immunodeficiency virus (HIV) 1 and 2, antibodies to Treponema pallidum antigens, hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus antigens at screening;
23. Positive result of rapid test for coronavirus disease pathogen 2019 (Coronavirus disease 2019, COVID-19) at screening;
24. Clinically significant electrocardiogram (ECG) abnormalities with a history and/or at screening;
25. Positive urinalysis for narcotics and potent drugs at screening;
26. Positive breath alcohol vapor test at screening;
27. Scheduling an inpatient stay during the study period, for any reason other than hospitalization required by this protocol;
28. Inability or inability to comply with the requirements of the protocol, to follow the procedures prescribed by the protocol, to observe the diet and activity regimen;
29. Vulnerable volunteer population: undergraduate and graduate medical, pharmacy, and dental students, clinical and laboratory assistants, pharmaceutical company employees, military personnel and prisoners, nursing home residents, low-income and unemployed persons, minorities, homeless, vagrants, refugees, persons in foster care, persons unable to consent, and law enforcement officers;
30. Other conditions that, in the opinion of the Investigator, would preclude the volunteer from being included in the study or could result in the early withdrawal of the volunteer from the study, including fasting or a special diet (e.g., vegetarian, vegan, salt restricted) or a special lifestyle (night work, extreme physical exertion).

Exclusion criteria:

1. Withdrawal of the volunteer from further participation in the study;
2. Failure of the volunteer to comply with the rules of participation in the study (skipping study procedures, independent use of drugs prohibited in the study, violation of dietary and lifestyle restrictions, etc.);
3. Causes/occurrence of situations during the study that jeopardize the safety of the volunteer (e.g. hypersensitivity reactions, etc.);
4. Volunteers selected for participation in the study in violation of the inclusion/non-inclusion criteria;
5. Development of serious/severe adverse event in a volunteer during the course of the study;
6. Volunteer is receiving or requires treatment that may affect the pharmacokinetics of the study drug;
7. Missing collection of 2 or more consecutive blood samples or 3 or more blood samples during a single Study Period;
8. Occurrence of vomiting/diarrhea within 6 h of administration of study drug;
9. Positive urine test for narcotics and potent drugs;
10. Positive breath alcohol vapor test;
11. A positive pregnancy test in women;
12. A positive test for COVID-19;
13. Occurrence of other reasons during the study that prevent the conduct of the study according to the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Maximum plasma concentration (Cmax) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - tmax | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Time to reach Cmax (tmax) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - AUC0-t | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - AUC0-inf | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - AUCextr | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Extrapolated AUC of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone, defined as (AUC0-inf - AUC0-t)/AUC0-inf
Pharmacokinetics - t1/2 | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Elimination half-life (t1/2) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - kel | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Elimination constant (kel) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - MRT | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Mean residence time (MRT) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - Vd | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Volume of distribution of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - CL | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  Clearance (CL) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - number of terminal timepoints | From 0 to 48 hours, (single dose); from 0 to 120 hours (multiple dose)
  number of points in the terminal logarithmic phase used to estimate the terminal elimination rate constant of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone

SECONDARY OUTCOMES:
Adverse event type | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  Adverse events will be assessed by complaints, results of physical examination, results of heart rate and blood pressure assessment, results of respiratory rate assessment, body temperature, laboratory monitoring (clinical blood count, biochemical blood count, urinalysis), electrocardiography; adverse events will be classified in accordance to MedDRA.
Adverse event frequency | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  Number and frequency of adverse events registered during the study
Adverse event severety | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  Severity of adverse events registered during the study
Drop-outs associated with adverse events | From Day -14 to Day -1 (screening), from Day 1 to Day 21 (single dosing and subsequent wash-out period), from Day 1 to Day 11 (multiple dosing and subsequent observation period)
  The number of cases of early termination of participation in the study due to the development of adverse events and/or serious adverse events associated with the study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Limited Liability Company "Medical Center Eco-Safety", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided